CLINICAL TRIAL: NCT03677973
Title: A Double-Blind, Randomized, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetic Profile of AB680 in Healthy Volunteers
Brief Title: A Study to Investigate the Safety of AB680 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB680CSP0001
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — quemliclustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: Dose Escalation (Active Comparator): Healthy volunteers will receive AB680 as a single intravenous (IV) infusion at 7 dose levels and as multiple IV infusions at 1 dose level. Assignment to receive AB680 or matching placebo will be random.
  Interventions: Drug: AB680
- Placebo: Dose Escalation (Placebo Comparator): Healthy volunteers will receive matching placebo as a single IV infusion and as multiple IV infusions. Assignment to receive AB680 or matching placebo will be random.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AB680 — AB680 is a Cluster of Differentiation (CD)73 Inhibitor
  Arms: Active: Dose Escalation
Other: Placebo — Matching Placebo
  Arms: Placebo: Dose Escalation

SUMMARY:
This is a double-blind, randomized, placebo-controlled, single- and multiple-ascending dose study to investigate the safety, tolerability, and pharmacokinetic profile of AB680 in healthy volunteers.

DETAILED DESCRIPTION:
AB680 will be administered as single and multiple intravenous doses to the healthy volunteers. In each group of 8 participants, 6 will receive AB680 and 2 will receive matching placebo.

The participants will be closely observed to monitor the general tolerability of AB680.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years, inclusive, at screening
* Body mass index 18 to 30 kg/m2
* Willing and able to sign informed consent
* Negative tests for hepatitis B surface antigen, anti-hepatitis C virus, and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening
* Healthy as determined by pre-study screening

Exclusion Criteria:

* History of clinically significant drug and/or food allergies
* Positive drug and alcohol screen at screening and (each) admission to the clinical research center.
* Participation in a drug study within 60 days prior to (the first) drug administration in the current study. Participation in more than 4 other drug studies in the 12 months prior to (the first) drug administration in the current study
* Participants who have significant infection or known inflammatory process on screening or admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs). | From First Dose Date to 15 Days After the Last Dose of AB680.
  Number of Participants with TEAEs as Assessed by CTCAE v5.0.
AB680 Peak Plasma Concentration (Cmax) | From First Dose Date to 15 Days After the Last Dose of AB680.
  Cmax as Measured by the Area Under Concentration-Time Curve from Plasma Collection and Analysis.
AB680 Time of Peak Concentration (Tmax) | From First Dose Date to 15 Days After the Last Dose of AB680.
  Tmax as Measured by the Time to Maximum Concentration-Time Curve from Plasma Collection and Analysis.

SECONDARY OUTCOMES:
Pharmacodynamic (PD) Effects of AB680 | From First Dose Date to 15 Days After the Last Dose of AB680.
  Enzymatic Activity of CD73 Measured in Participant Blood Samples.
Plasma Levels of Adenosine | From First Dose Date to 15 Days After the Last Dose of AB680.
  Amount of Adenosine Measured in Participant Blood Samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Melbourne, VIC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- [Derived] Bowman CE, da Silva RG, Pham A, Young SW. An Exceptionally Potent Inhibitor of Human CD73. Biochemistry. 2019 Aug 6;58(31):3331-3334. doi: 10.1021/acs.biochem.9b00448. Epub 2019 Jul 23. PMID 31334635
- See also: AB680CSP0001 - Lay Summary (English Version) — https://trials.arcusbio.com/study/?id=AB680CSP0001